CLINICAL TRIAL: NCT04712851
Title: A Phase II Open-Label, Single Arm Pilot Study to Evaluate the Safety and Efficacy of Pembrolizumab for High-Grade Cervical Intraepithelial Neoplasia
Brief Title: Pembrolizumab for the Treatment of Cervical Intraepithelial Neoplasia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-002121; NCI-2020-11457 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-01-12; First posted 2021-01-15 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Cervical Intraepithelial Neoplasia; Cervical Squamous Cell Carcinoma In Situ; Cervical Squamous Intraepithelial Neoplasia 2
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (pembrolizumab) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 6 weeks for 4 cycles (24 weeks).
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase II trial studies the effect of pembrolizumab on cervical intraepithelial neoplasia. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Proportion of subjects with pathologic complete response (no evidence of dysplasia).

SECONDARY OBJECTIVES:

I. Safety and tolerability of pembrolizumab in subjects with cervical intraepithelial neoplasia (CIN).

II. Proportion of subjects with pathologic partial response (regression to a lower grade of dysplasia).

EXPLORATORY OBJECTIVES:

I. Evaluation of Programmed Death-Ligand 1 (PD-L1) expression in CIN lesions as a biomarker of response to therapy.

II. Evaluation of Human Papillomavirus (HPV) status as a biomarker of response to therapy.

III. Evaluation of HPV clearance as a surrogate endpoint.

OUTLINE:

Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Treatment repeats every 6 weeks for 4 cycles (24 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Female participants who are at least 21 years of age on the day of signing informed consent with active (not yet resected), histologically confirmed diagnosis of CIN grade 2 or 3 or carcinoma in situ (without invasive component) will be enrolled in this study. Subjects with multifocal disease are acceptable
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP) OR
  * A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 120 days after the last dose of study treatment
* The participant (or legally acceptable representative if applicable) provides written informed consent for the trial
* Have provided archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue
* Participants must be willing to consent to mid-study biopsy after cycle 2 of treatment if there is an accessible lesion and biopsy is not contraindicated
* Participants must be willing to consent to either loop electrode excision procedure (LEEP) or cold-knife cone (CKC) at the end of treatment (i.e., after 24 weeks on study), unless surgery is contraindicated at that time
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Have normal organ function (with all baseline laboratory assessments in the normal range). Specimens must be collected within 10 days prior to the start of study treatment, except for pregnancy test which must be within 72 hours of cycle 1 of treatment

Exclusion Criteria:

* A WOCBP who has a positive urine pregnancy test within 72 hours prior to allocation. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

  * Note: in the event that 72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative in order for subject to start receiving study medication
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137)
* Has received prior systemic therapy for CIN including investigational agents within the prior 4 weeks [could consider shorter interval for short half-life drugs] prior to allocation.

  * Note: Participants must have recovered from all adverse events (AEs) due to previous therapies to =< grade 1 or baseline. Participants with =< grade 2 neuropathy may be eligible.
  * Note: If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment
* Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (=< 2 weeks of radiotherapy) to non-central nervous system (CNS) disease
* Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guerin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist) are live attenuated vaccines and are not allowed
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.

  * Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug
* Has a history of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years.

  * Note: The time requirement does not apply to participants who underwent successful definitive resection of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, in situ cervical cancer, or other in-situ cancers
* Has severe hypersensitivity (>= grade 3) to pembrolizumab and/or any of its excipients
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis
* Has an active infection requiring systemic therapy
* Has a known history of human immunodeficiency virus (HIV) infection

  * Note: No HIV testing is required unless mandated by local health authority
* Has a known history of hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or known active hepatitis C virus (defined as HCV ribonucleic acid [RNA] [qualitative] is detected) infection. Note: no testing for hepatitis B and hepatitis C is required unless mandated by local health authority
* Has a known history of active TB (Bacillus tuberculosis)
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment
* Has had an allogenic tissue/solid organ transplant

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Pathological response rate | At 6 months
  Will assess the percent of patients with pathologic complete response at 6 months.

SECONDARY OUTCOMES:
Proportion of subjects with pathologic partial response (regression to a lower grade of dysplasia) | Up to 6 months
Incidence of adverse events | Up to 6 months

OTHER OUTCOMES:
PD-L1 expression | Up to 6 months
  Will correlate PD-L1 positivity with response to pembrolizumab.
Assess percentage of subjects who respond to treatment who are HPV positive compared to percentage of subjects who respond to treatment who are HPV negative. | Up to 6 months
  Assess percentage of subjects who respond to treatment who are HPV positive (using p16 positivity from pathology) compared to percentage of subjects who respond to treatment who are HPV negative in order to evaluate if HPV positivity correlates with improved response to treatment.
Assess percentage of subjects with initial HPV infection who clear HPV infection (using p16 positivity from pathology) as a surrogate response to treatment evaluation. | Up to 6 months
  Will evaluate HPV clearance as a surrogate endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: John A Glaspy, MD, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- University of California at Los Angeles / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States